CLINICAL TRIAL: NCT02454153
Title: Hyperglycemic Profiles in Obstructive Sleep Apnea: Effects of PAP Therapy
Acronym: HYPNOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00093188; R01HL117167 (NIH)
Record Dates: First submitted 2015-01-14; First posted 2015-05-27 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Sleep Apnea; Diabetes
MeSH Terms: conditions — Sleep Apnea Syndromes; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- REMStar Positive Airway Pressure (Active Comparator): Positive pressure therapy is the standard of care for managing obstructive sleep apnea.
  Interventions: Device: REMStar Positive Airway Pressure
- LifeStyle Counseling (Other): Lifestyle guidelines developed by the American Diabetes Association for weight loss will be provided to all subjects.
  Interventions: Behavioral: LifeStyle Counseling

INTERVENTIONS:
Device: REMStar Positive Airway Pressure — Positive airway pressure therapy is the standard of care for managing obstructive sleep apnea
  Arms: REMStar Positive Airway Pressure
Behavioral: LifeStyle Counseling — Lifestyle guidelines developed by the American Diabetes Association for weight loss will be provided to all subjects.
  Arms: LifeStyle Counseling

SUMMARY:
This is a randomized control trial in people with diabetes and obstructive sleep apnea who will be randomly assigned for 3 months to PAP therapy along with healthy lifestyle and sleep education or healthy lifestyle and sleep education.

DETAILED DESCRIPTION:
Research over the last decade has shown that obstructive sleep apnea (OSA) is a common condition in people with diabetes. Observational and experimental evidence also indicates that intermittent hypoxemia and recurrent arousals in OSA may alter glucose metabolism and worsen glycemic control. However, the impact of treating OSA with positive airway pressure (PAP) therapy on glycemic variability and control is not well defined. Adequately powered randomized clinical trials have yet to be performed to demonstrate whether PAP therapy for OSA in diabetics can improve glycemic variability (and control), decrease blood pressure, and reverse endothelial dysfunction. The overarching goal of this study is to determine whether PAP therapy for OSA in diabetics leads to improvements in (a) glycemic variability as assessed by self-monitoring of blood glucose and continuous monitoring of glucose; (b) glycosylated hemoglobin; (c) blood pressure; (d) endothelial function; (e) serum and urinary biomarkers; and (f) dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics
* Age > 21 and ≤ 75 years

Exclusion Criteria:

* Inability to consent or commit to the required visits
* Use of insulin or other injections for diabetes
* Weight change of 10% in last six months
* Use of oral steroids in the last six months
* Pulmonary disease (i.e., COPD)
* Renal or hepatic insufficiency
* Recent MI or stroke (< 3 months)
* Sleep-related hypoventilation
* Obesity-hypoventilation syndrome
* Morbid Obesity
* Occupation as a commercial driver or operator of heavy machinery
* Active substance use
* Untreated thyroid disease
* Pregnancy
* Any history of seizures or other neurologic disease
* Poor sleep hygiene or sleep disorder other than sleep apnea
* Central sleep apnea
* Variants of obstructive sleep apnea (e.g., REM-related OSA)
* Participants not suitable for the study based on the clinical judgment
* Use of any investigational drug within the past 30 days
* Participating in another study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naresh M Punjabi, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Aurora RN, Rooney MR, Wang D, Selvin E, Punjabi NM. Effects of Positive Airway Pressure Therapy on Glycemic Variability in Patients With Type 2 Diabetes and OSA: A Randomized Controlled Trial. Chest. 2023 Oct;164(4):1057-1067. doi: 10.1016/j.chest.2023.04.017. Epub 2023 Apr 14. PMID 37062349
- [Derived] Fang M, Wang D, Rooney MR, Echouffo-Tcheugui JB, Coresh J, Aurora RN, Punjabi NM, Selvin E. Performance of the Glucose Management Indicator (GMI) in Type 2 Diabetes. Clin Chem. 2023 Apr 3;69(4):422-428. doi: 10.1093/clinchem/hvac210. PMID 36738249
- [Derived] Selvin E, Wang D, Rooney MR, Fang M, Echouffo-Tcheugui JB, Zeger S, Sartini J, Tang O, Coresh J, Nisha Aurora R, Punjabi NM. Within-Person and Between-Sensor Variability in Continuous Glucose Monitoring Metrics. Clin Chem. 2023 Feb 1;69(2):180-188. doi: 10.1093/clinchem/hvac192. PMID 36495162
- [Derived] Selvin E, Wang D, Rooney MR, Echouffo-Tcheugui J, Fang M, Zeger S, Sartini J, Tang O, Coresh J, Aurora RN, Punjabi NM. The Associations of Mean Glucose and Time in Range from Continuous Glucose Monitoring with HbA1c in Adults with Type 2 Diabetes. Diabetes Technol Ther. 2023 Jan;25(1):86-90. doi: 10.1089/dia.2022.0178. Epub 2022 Nov 23. PMID 36108310
- [Derived] Rooney MR, Aurora RN, Wang D, Selvin E, Punjabi NM. Rationale and design of the Hyperglycemic Profiles in Obstructive Sleep Apnea (HYPNOS) trial. Contemp Clin Trials. 2021 Feb;101:106248. doi: 10.1016/j.cct.2020.106248. Epub 2020 Dec 11. PMID 33316455

RESULTS

PARTICIPANT FLOW:
Groups:
- REMStar Positive Airway Pressure: Positive pressure therapy is the standard of care for managing obstructive sleep apnea. Participants also received Lifestyle counseling as described below.
  REMStar Positive Airway Pressure: Positive airway pressure therapy is the standard of care for managing obstructive sleep apnea
  Lifestyle guidelines developed by the American Diabetes Association for weight loss will be provided to all subjects.
  LifeStyle Counseling: Lifestyle guidelines developed by the American Diabetes Association for weight loss will be provided to all subjects.
Period: Overall Study
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Started | 92 | 92
Completed | 92 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (8.6) | 60.8 (9.6) | 59.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 50 | 90
  Male | 52 | 42 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 34 | 63
  White | 53 | 50 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.8 (5.5) | 33.7 (5.8) | 33.8 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Continuous Glucose Monitoring System Standard Deviation
Description: Continuous Glucose Monitoring Metrics - change in standard deviation between baseline and three months.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 92 | 92
mg/dL | 0.8 (6.7) | 1.1 (8.6)

2. Secondary Outcome: Mean Difference in Systolic Blood Pressure
Description: Mean difference between 3 months and baseline systolic blood pressures (in mmHg) by group.
Time Frame: Baseline and 3 months
Population: Missing data is due to participants who did not have their blood pressure taken at three month timepoint.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 87 | 88
mmHg | -7.3 (6.1) | 7.4 (5.8)

3. Secondary Outcome: Change in Endothelial Dysfunction as Assessed by the Reactive Hyperemic Index
Description: Endothelial function was measured by the EndoPAT device - difference at 3 months - baseline, by group. The outcome reported is the Reactive Hyperemic Index (RHI). The RHI is a measure of endothelial vasodilator function. The RHI is the post-to-pre occlusion peripheral arterial tone signal ratio in the occluded arm relative to the other arm, which is not occluded. Persons with worse endothelial function have a lower RHI score. Consequently, a low RHI indicates more endothelial dysfunction. A value of 1.67 or less is considered abnormal vascular tone. The reported lower and upper limits in adults with type 2 diabetes is 1.1 - 4.9.
Time Frame: Baseline and 3 months
Population: Missing data is due to participants who did not complete the procedure at three months.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- REMStar Positive Airway Pressure: Positive pressure therapy is the standard of care for managing obstructive sleep apnea.
  REMStar Positive Airway Pressure: Positive airway pressure therapy is the standard of care for managing obstructive sleep apnea.
  Lifestyle guidelines developed by the American Diabetes Association for weight loss will be provided to all subjects.
  LifeStyle Counseling: Lifestyle guidelines developed by the American Diabetes Association for weight loss will be provided to all subjects.
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 86 | 85
ratio | -0.0014 (0.65) | 0.0024 (0.69)

4. Secondary Outcome: Heart Rate Variability
Time Frame: 3 months
Population: No data was collected
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in the Epworth Sleepiness Scale
Description: The Epworth Sleepiness Scale measures self-reported sleep propensity or daytime sleepiness. The range of the scale is 0 to 24 (integers only), with increasing values corresponding to increasing sleepiness. A cut-point of ≥ 11 is also sometimes used to differentiate those with pathological sleepiness (≥ 11) versus those without < 11. The difference between the three month final visit - the baseline visit score is reported by group
Time Frame: Baseline and 3 months
Population: Missing data points were due to participants not completing the survey at three months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 83 | 83
units on a scale | -2.5 (4.3) | -1.3 (3.1)

6. Secondary Outcome: Change in Post-Pre Meal Blood Glucose Levels
Description: The difference from baseline to three months in self-reported in blood glucose levels before and after meals (mg/dL) (post-meal - pre-meal). Data is presented for breakfast, lunch, and dinner.
Time Frame: Baseline and 3 months
Population: One participant in the REMStar Positive Airway Pressure arm was missing data on the three month visit.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 91 | 92
mg/dL
  Change post-pre breakfast | -9.9 (4.8) | -1.3 (4.8)
  Change post-pre lunch | 1.0 (5.4) | -6.1 (5.4)
  Change post-pre dinner | -3.0 (5.1) | 3.7 (5.1)

7. Secondary Outcome: Change in Glycosylated Hemoglobin A1c Level
Description: Change in point-of-care hemoglobin A1c (%) after three months.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 92 | 92
percentage of glycosylated hemoglobin | 0.2 (0.7) | 0.2 (0.9)

8. Secondary Outcome: Continuous Glucose Monitoring System Mean Amplitude Glucose Excursion
Description: Mean Amplitude Glucose Excursion in mg/dL (difference between the peaks and troughs of glucose from continuous glucose monitoring at three months).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 92 | 92
mg/dL | 69.5 (20.5) | 71.4 (20.4)

9. Secondary Outcome: Continuous Glucose Monitoring System Standard Deviation
Description: The standard deviation of the glucose from continuous glucose monitoring at three months.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 92 | 92
mg/dL | 38.7 (11.3) | 39.2 (10.8)

10. Secondary Outcome: Change in Continuous Glucose Monitoring System Mean Glucose
Description: Continuous Glucose Monitoring Metric - change in average glucose level (mg/dL) from baseline to three months.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
Number analyzed (Participants) | 92 | 92
mg/dL | 4.3 (25.3) | 9.5 (29.3)

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | REMStar Positive Airway Pressure | LifeStyle Counseling
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 1/92 | 0/92
Other Adverse Events (participants affected / at risk) | 0/92 | 0/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REMStar Positive Airway Pressure (N=92) | LifeStyle Counseling (N=92)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — Hospital admission for a right-sided stroke. Event reported to the Institutional Review Board and deemed not to be related to the research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT02454153/Prot_SAP_000.pdf